CLINICAL TRIAL: NCT03143439
Title: Evaluation of the Fathers Advancing Communities Together (FACT) Program
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Urban Institute (Other)
Collaborators: Rubicon Programs (Unknown)
Responsible Party: Principal Investigator, Lindsey Cramer, Research Associate, Urban Institute
Other Study IDs: 09226-000-00
Record Dates: First submitted 2017-03-30; First posted 2017-05-08 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Responsible Fatherhood Programming

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Program group: The program group will be comprised of all individuals who enrolled in the FACT program from July 2016 through September 2019 and have active child support cases with the Contra Costa County Department of Child Support Services.
  Interventions: Behavioral: Fathers Advancing Communities Together (FACT) program
- Comparison group: The comparison group will be comprised of individuals with active child support cases with the Contra Costa County Department of Child Support Services who are demographically comparable to the treatment group (i.e., FACT fathers with active child support cases), yet did not participate in or receive FACT services.

INTERVENTIONS:
Behavioral: Fathers Advancing Communities Together (FACT) program — The FACT program offers fathers and their families responsible parenting, healthy relationship, and economic stability services and activities.
  Groups: Program group

SUMMARY:
The Urban Institute-a nonprofit, nonpartisan research organization-is partnering with Rubicon Programs to conduct a rigorous evaluation of its Fathers Advancing Communities Together (FACT) program. FACT is a multi-faceted program designed to deliver responsible parenting, healthy relationships, and economic stability services on a voluntary basis to low-income fathers in Contra Costa County, California. Urban's evaluation comprised of three key components:

The implementation evaluation will describe FACT program activities and services, including communication and coordination across partners, service delivery mechanisms, and whether and how participants and their families received comprehensive services. Urban will identify a logic model for the program and assess the barriers to and facilitators of program performance. The implementation evaluation will draw from interviews with program staff, partners, and stakeholders, as well as field observations, program and administrative data, and focus groups with FACT participants and their families.

The outcome evaluation will build on the implementation evaluation to determine whether specific program components, their frequency, and their duration, are related to outcomes. Urban will conduct surveys of program participants at the time of their enrollment into the program and one year following their enrollment to explore how participants' self-reported attitudes on various domains are associated with economic self-sufficiency and family functioning. Urban will also use program and administrative data collected by Rubicon and its partners, specifically Rubicon's case management database, to assess participant outcomes.

The impact evaluation will assess to what extent participation in the FACT program is associated with improved outcomes as compared to similarly situated individuals who did not participate in the program. Urban will work with Rubicon's partners to identify individuals living in Contra Costa County who were eligible to participate in the program but, for whatever reason, did not do so. Once a comparison group of fathers has been established, Urban will use individual-level outcome data to determine whether the FACT program has an impact on economic self-sufficiency and family functioning.

ELIGIBILITY:
Inclusion Criteria:

* An individual is eligible for the impact evaluation if the individual is a FACT participant and is a parent with an open child support case in Contra Costa County, CA during the time of their enrollment.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: The study population will include all FACT participants enrolled from July 2016 through September 2019. An individual is eligible to enroll in FACT if the individual is a parent with a child under 18, classified as having low income, lives in Contra Costa County, and is interested in services to enhance financial mobility. The participant survey will be administered to a sub-sample of approximately 200-250 FACT participants enrolled from March 2017 to March 2019. The sub-sample for the impact evaluation will be FACT participants with an active child support case.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-09-30 (Actual); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Increases in child support payment modifications | 6 months
  The outcome is a dichotomous measure of whether the individual had any child support modifications between enrollment and 6-months post enrollment (1 = Yes; 0 = No).
Increases in monthly child support payment amounts | 6 months
  This outcome is a semi-continuous measure indicating the average dollar amount of monthly child support payments between enrollment and 6-months post enrollment in dollars
Increases in employment | 6 months
  This outcome is a dichotomous measure of whether the individual was employed at any point between enrollment and 6-months post enrollment (1 = Yes; 0 = No).
Increases in receipt of public assistance | 6 months
  This outcome is a dichotomous measure of whether an individual was on any public assistance (e.g., TANF and SNAP) at any point between enrollment and 6-months post enrollment (1 = Yes; 0 = No).

SECONDARY OUTCOMES:
Court orders | 6 months
  The outcome is a dichotomous measure of whether there was a new child support court order during the 6-month period after enrollment (1 = Yes; 0 = No).
Amount of court orders | 6 months
  This outcome is a semi-continuous measure indicating the total dollar amounts of new court orders during the 6-month period after enrollment.
Arrear | 6 months
  This outcome is a dichotomous measure of whether there was a new arrear (an open case with unpaid child support owed to the custodial parent) at 6-months post enrollment.
Arrear balance | 6 monhts
  This outcome is a semi-continuous measure of the total balance of new arrears at 6-months post enrollment.
Months on public assistance | 6 months
  This outcome measure is a count of the number of months individuals were on any public assistance during the 6-month period after enrollment.

OTHER OUTCOMES:
Improvement in fathers' attitudes and perceptions of economic self-sufficiency, relationships, and parenting as measured by participant-level surveys, program data, and administrative data. | One year (baseline and one-year follow up)
  This outcome will capture how, due to FACT programming, participants' changes in attitudes and perceptions of their parenting, relationships, and economic stability were associated with changes in program-specific behaviors/outcomes, and the extent to which program components (e.g., classes and workshops) were associated with changes in fathers' attitudes, perceptions, and behaviors as measured by a participant survey. This outcome will draw on data collected from participant surveys, program data in Rubicon's Salesforce/ECM database, and administrative data from Rubicon's partners providing services to FACT participants. All of the above data points will be combined and linked, to the extent possible, to analyze individual-level data to assess participants' changes in their attitudes and perceptions of self-sufficiency, relationships, and parenting.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Cramer, Principal Investigator — Urban Institute; Bryce Peterson, PhD, Principal Investigator — Urban Institute
Locations (1):
- Rubicon Programs, Richmond, California, United States